CLINICAL TRIAL: NCT06937762
Title: Intracapsular Coblation Tonsillotomy Versus Extracapsular Radiofrequency and Cold Knife Dissection Tonsillectomy
Brief Title: Coblation Tonsillotomy Versus Radiofrequency and Cold Knife Dissection Tonsillectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Magdi Noaman Othman Orabi, Principal Investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KFSIRB200-561
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Tonsillitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intra capsular coblation tonsillotomy (Active Comparator)
  Interventions: Device: Intra capsular coblation tonsillotomy
- Extracapsular cold knife dissection tonsillectomy (Active Comparator)
  Interventions: Device: Extracapsular cold knife dissection tonsillectomy
- Extra capsular Radiofrequency tonsillectomy (Active Comparator)
  Interventions: Device: Extra capsular Radiofrequency tonsillectomy

INTERVENTIONS:
Device: Intra capsular coblation tonsillotomy — Tonsils were dissected from the surface inward with the wand set at Coblate 7 setting. The wand skims the tonsil surface with continuous saline irrigation. Ablation was performed without penetrating the tonsillar capsule. Retraction of the tonsillar pillars is done to define the margins for near complete ablation. When the capsule is approached, the wand is turned down to Coblate 3 setting. Thin layer of tonsillar tissue is left to protect the capsule. Bleeding does not occur in most cases, but when it occurs, the wand was used in the Coagulate 5 setting for homeostasis
  Arms: Intra capsular coblation tonsillotomy
Device: Extracapsular cold knife dissection tonsillectomy — Begin by retracting the anterior tonsillar pillar to expose the tonsil, use a cold knife (scalpel or tonsil dissector) to make an incision along the anterior pillar near the mucosal margin of the tonsil, identify the plane between the tonsillar capsule and the underlying pharyngeal muscle, then carefully dissect the tonsil away from the surrounding tissues, following the plane to avoid trauma to the underlying structures, proceed from the superior pole of the tonsil to the inferior pole, ensuring that the entire tonsil is removed, use gauze or sponges to control minor bleeding during the procedure, for more significant bleeding, apply direct pressure or use ligatures and cold packs, achieve final hemostasis using absorbable sutures or electrocautery if needed
  Arms: Extracapsular cold knife dissection tonsillectomy
Device: Extra capsular Radiofrequency tonsillectomy — Radiofrequency bipolar forceps, connected to a radiofrequency apparatus model Ellman Surgitron 4 MHz (Ellman International, New York, USA) by which cutting and dissection with coagulation were done in the same time with minimal diffuse heating to the surrounding tissue. The power was adjusted to a power grade 40 in a bipolar mode.
  Arms: Extra capsular Radiofrequency tonsillectomy

SUMMARY:
This study aims to assess and compare the outcomes between coblation intracapsular tonsillotomy versus extracapsular Radiofrequency and cold knife dissection tonsillectomy efficacy in managing patients requiring tonsil surgery as regards (time of operation, Intraoperative blood loss, postoperative pain, postoperative bleeding, complications, tonsillar fossa healing)

ELIGIBILITY:
Inclusion criteria:

Recurrent Acute tonsillitis Tonsillitis resulting in febrile convulsions Enlarged tonsils that cause upper airway obstruction, dysphagia, sleep disorders Chronic tonsillitis Chronic or recurrent tonsillitis in a streptococcal carrier not responding to beta-lactamase-resistant antibiotics

Exclusion criteria:

Patients with known bleeding disorders Acute infections of tonsil Contraindications for general anesthesia Anemia Patients unwilling or unable to give informed consent were excluded from this study patients

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
comparision of the severity of postoperative pain between the three groups. | The first time on day 1, the second time on day 3 and third time on day 7
  1- Postoperative pain will be assessed using visual analogue scale (VAS) from 0 (no pain) to 10 (worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University Hospitals, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Metcalfe C, Muzaffar J, Daultrey C, Coulson C. Coblation tonsillectomy: a systematic review and descriptive analysis. Eur Arch Otorhinolaryngol. 2017 Jun;274(6):2637-2647. doi: 10.1007/s00405-017-4529-4. Epub 2017 Mar 18. PMID 28315933
- [Background] Liu Q, Zhang Y, Lyu Y. Postoperative hemorrhage following coblation tonsillectomy with and without suture: A randomized study in Chinese adults. Am J Otolaryngol. 2021 Jan-Feb;42(1):102760. doi: 10.1016/j.amjoto.2020.102760. Epub 2020 Oct 18. PMID 33125902